CLINICAL TRIAL: NCT06666569
Title: Evaluation of the Effectiveness of Kits Promonitor-IFX/ADL and Promonitor-Anti-IFX/ADL to Assist in Taking Clinical Decisions in Patients With IBD Treated With IFX or ADA
Brief Title: Evaluation of the Effectiveness of Kits Promonitor-IFX/ADL and Promonitor-Anti-IFX/ADL in Patients With IBD
Acronym: IBDMonitor
Status: Completed | Type: Observational
Sponsor: Hospital de Basurto (Other)
Collaborators: PROGENIKA BIOPHARMA, A GRIFOLS Company (Unknown)
Responsible Party: Principal Investigator, Maria del Carmen Muñoz Villafranca, Principal Investigator, Hospital de Basurto
Other Study IDs: IBD-MONITOR
Record Dates: First submitted 2024-10-24; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Crohn Disease and Ulcerative Colitis
Keywords: IBD, Anti-TNFα, Promonitor-IFX/ADL, Promonitor-Anti-IFX/ADL
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 32 Months
Biospecimen Retention: Samples Without DNA — Leftover serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention Cohort and Clinical Practice Cohort: Cohort of routine practice, where the clinician will be blinded to these results.
  The randomization process will be by blocks and weighted to the ADL/IFX ratio of use of these treatments in the usual clinical practice of the participating hospitals, to guarantee a homogeneous distribution of the treatments in the groups at the beginning/end of the follow-up.
  Interventions: Device: Use of the test for treatment optimization

INTERVENTIONS:
Device: Use of the test for treatment optimization — Intervention cohort, where the clinician will have information on the test results to support decision making on treatment optimization. The randomization process will be by blocks and weighted to the ADL/IFX ratio of use of these treatments in the usual clinical practice of the participating hospitals, to guarantee a homogeneous distribution of the treatments in the groups at the beginning/end of the follow-up.

SUMMARY:
To establish the efficacy, safety, effectiveness and efficiency of monitoring the levels of anti-TNFα drugs and the levels of antibodies generated against these drugs in the treatment of patients with moderate or severe IBD (CD/CU).

An analysis will be made of the economic impact on the Health System of monitoring treatment with anti-TNFα drugs in CD/CU.

As a result of this specific objective, a standardized procedure will be established for the evaluation of the response to treatment with anti-TNFα drugs for CD/CU that includes the new trials and the new devices developed.

DETAILED DESCRIPTION:
* To evaluate whether a dose and plasma level optimization strategy based on the use of Promonitor-IFX, Promonitor-Anti-IFX, Promonitor-ADL, and Promonitor-Anti-ADL kits in CD/CU patients on IFX/ADL treatment is superior in terms of the percentage of patients in clinical remission at 12 months compared to standard practice.
* To evaluate whether a dose and plasma level optimization strategy based on the use of Promonitor-IFX, Promonitor-Anti-IFX, Promonitor-ADL, and Promonitor-Anti-ADL kits in CD/CU patients on IFX/ADL treatment is superior in terms of the percentage of patients in deep remission at 12 months compared to standard practice.
* To analyze the influence of the use of the IFX/ADL antibody detection test in moderate to severe CD/CU patients on the annual direct cost to the health system of these patients, compared to the non-use of the tests.
* To evaluate the effectiveness of IFX/ADL antibody testing in moderate to severe CD/CU patients on the increase in quality-adjusted life-years compared to non-use of the tests.
* To evaluate the effectiveness of testing for antibodies to IFX/ADL in moderate to severe CD/CU patients in reducing the number of flares, compared to not using the tests.

Exploratory objective - To conduct a cost-effectiveness (utility) analysis of a strategy for the management of stable moderate to severe CD/CU patients based on treatment monitoring.

Page 10 of 83 anti-TNFα with the introduction of screening tests for plasma levels/antibodies to IFX/ADL with respect to standard practice based on clinical signs/symptoms.

Main operational objective

- To assess whether the prevalence of 1-year remission in moderate to severe CD/CU patients whose anti-TNFα treatment has been managed using Promonitor IFX/ADL kits is at least 16% higher compared to the group of patients in whom this technique has not been employed.

ELIGIBILITY:
Inclusion criteria:

* patients of both sexes
* over 18 years of age
* diagnosis of CD/CU confirmed by endoscopy
* stable clinical status (remission) for at least 12 weeks prior to inclusion in the study
* on treatment with IFX/ADL for at least 3 months with stabilized dosage and outside the induction period
* negative for tuberculosis at the start of treatment
* who sign the informed consent form

Exclusion criteria:

* severe concomitant pathology preventing adequate follow-up of patients.
* continued corticosteroid therapy at prednisone equivalent doses higher than 40 mg/day
* patients with positive antibody levels at baseline
* there is treatment with immunomodulators and/or corticoids, when it is at high doses and with variations in time
* Patients with intestinal resection and Crohn's disease in prophylactic treatment with anti-TNF, but without recurrence.
* who are participating in a clinical trial or interventional study. Participation in the study will be offered to all patients who meet the above criteria, and in a consecutive manner, without a prior selection process. The comparison group will consist of a cohort of patients belonging to the same Digestive Services and meeting the same selection criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease (Crohn's disease or ulcerative colitis) on treatment with Infliximab or Adalimumab and who have been clinically stable for 12 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Pharmacological management of IBD | 32 meses
  Follow-up of two cohorts made up of patients diagnosed with moderate severe CD/UC, from the Basurto University Hospital, Cruces University Hospital and San Eloy Hospital, and who are being treated with IFX/ADL, and stable in terms of disease activity

CONTACTS AND LOCATIONS:
Locations (1):
- Basurto University Hospital, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR